CLINICAL TRIAL: NCT03356158
Title: A Phase 1 Study of Recombinant Anti-Epidermal Growth Factor Receptor (EGFR) Human-mouse Chimeric Monoclonal Antibody Injection in Patients With Metastatic Colorectal Cancer
Brief Title: A Study of Recombinant Anti-EGFR Monoclonal Antibody in Patients With Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPGJ602-001
Record Dates: First submitted 2017-11-09; First posted 2017-11-29 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2017-11

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic Colorectal Cancer,; Recombinant Anti-EGFR Monoclonal Antibody
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CPGJ 602 low dose (Experimental): Part 1: CPGJ602, IV over 2 hours, 100 mg/m2 X 1;
  Interventions: Biological: CPGJ602
- CPGJ 602 normal dose (Experimental): Part 1: CPGJ602, IV over 2 hours, 400 mg/m2 X 1; Part 2: CPGJ602, IV, QW, 400 mg/m2 X 1, over 2 hours, followed by 250mg/m2 X4, over 1 hour for each time;
  Interventions: Biological: CPGJ602
- Cetuximab normal dose (Active Comparator): Part 1: Cetuximab, IV over 2 hours, 400 mg/m2 X 1. Part 2: Cetuximab, IV, QW, 400 mg/m2 X 1, over 2 hours, followed by 250mg/m2 X4, over 1 hour for each time.
  Interventions: Biological: Cetuximab

INTERVENTIONS:
Biological: CPGJ602 — Injection, q.w., 20 mg: 100 ml
  Arms: CPGJ 602 low dose; CPGJ 602 normal dose
Biological: Cetuximab — Injection, q.w., 20 mg: 100 ml
  Arms: Cetuximab normal dose

SUMMARY:
This is an open-label, parallel designed study to assess the pharmacokinetics, safety and tolerability of the single-dose and multi-dose of a recombinant anti-EGFR monoclonal antibody (CPGJ602) in patients with at least one prior chemical regimen failed metastatic colorectal cancer. The immunogenicity and preliminary efficacy of CPGJ602 will also be assessed. The study includes 3 parts: part 1: after a single dose of CPGJ602 or cetuximab (the active comparator), the patients will be observed for 4 weeks; part 2: CPGJ602 or cetuximab will be administered to the patients once a week for 5 weeks; part 3: CPGJ602 will be administered to the patients once a week until the patient's death or the withdrawal decision of the patient and/or investigator.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary:

To assess the pharmacokinetics, safety and tolerability of the single-dose and multi-dose of CPGJ602 administered by intravenous infusion.

Secondary:

To assess the immunogenicity and anti-tumor activity of CPGJ602, compare the pharmacokinetics and immunogenicity between CPGJ602 and the active comparator, cetuximab, and to provide scientific basis for the subsequent phase 2/3 clinical trials.

OUTLINE:

This is an open-label, parallel designed study in patients with at least one prior chemical regimen failed metastatic colorectal cancer. The study can be divided into 3 parts:

Part 1: Single-dose Part

* Arm A: CPGJ602, IV over 2 hours, 100 mg/m2 X 1;
* Arm B: CPGJ602, IV over 2 hours, 400 mg/m2 X 1;
* Arm C: Cetuximab, IV over 2 hours, 400 mg/m2 X 1.

Part 2: Multi-dose Part

The subjects from arm A in Part 1 will be randomized into arm B or C.

* Arm B: CPGJ602, IV, QW, 400 mg/m2 X 1, over 2 hours, followed by 250mg/m2 X4, over 1 hour for each time;
* Arm C: Cetuximab, IV, QW, 400 mg/m2 X 1, over 2 hours, followed by 250mg/m2 X4, over 1 hour for each time. The completion of Day 63 Visit (the visit on the 7th day after the 5th dose in Part 2) can be considered as the completion of the study.

Part 3 (Follow-up Part)

CPGJ602, IV over 1 hour, QW, 250mg/m2, until the patient's death or the withdrawal decision of the patient and/or investigator.

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years old, male or female.
2. Histologically or cytologically confirmed metastatic CRC, and have failed (disease progression or intolerance) at least one prior chemical regimen containing oxaliplatin, irinotecan or 5-FU, etc.
3. ECOG performance status 0 or 1.
4. Estimated life expectancy ≥ 3 months.
5. RAS (including K-ras and N-ras) wide type status.
6. Adequate bone marrow, hepatic and renal functions. Hematopoietic:

   Leukocytes (WBC)>4.0×109/L or Absolute Neutrophil Count (ANC)> 1.5×109/L, Platelet Count (PLT)>80×109/L, Hemoglobin (Hb)>90g/ L; Hepatic: Total Bilirubin (T-Bil)≤1.5×ULT (Upper Limit of Normal), Alanine Transaminase (ALT)/ Aspartate Transaminase (AST)≤2.5×ULT or ≤5×ULT in case of liver metastases; Renal: Blood Urea Nitrogen (BUN)≤1.5×ULT, Serum Creatinine (Cr) ≤ 1.5×ULT.
7. At least one measurable disease based on RECIST criteria (v 1.1).
8. Signed informed consent on a voluntary basis at screening, and no geographical condition that would preclude the study compliance.

Exclusion Criteria:

1. Less than 28 days since prior chemotherapy, radiotherapy or surgery (diagnosis biopsy is allowed).
2. Previous epidermal growth factor receptor (EGFR) targeted therapies (including monoclonal antibody, tyrosine kinase inhibitor [TKI] and other EGFR targeted therapies, such as cetuximab, nimotuzumab, panitumumab, gefitinib, erlotinib, and icotinib, etc.
3. Known hypersensitivity to study drugs or any of the excipients.
4. Known or clinical suspected brain metastases and/or disease of meninges.
5. Clinically significant cardiovascular or cerebrovascular dis ease, history of myocardial infarction (MI) in the latest 6 months, or high-risk of uncontrolled cardiac arrhythmias.
6. History of acute or sub-acute intestinal obstruction, or of inflammatory bowel disease.
7. A serious and uncontrolled concomitant disease which, in the investigator's opinion, rules out the patient's participation in the study, such as history of malignancies other than CRC (with the exception of: curatively treated carcinoma of the skin [except for melanoma]; cured cervical cancer or basal cell skin cancer, ductal carcinoma in situ [DICS], endometrial carcinoma [stage I grade 1]; and other solid tumors including lymphoma without bone marrow infiltration for which the patient has been disease-free for 5 years), uncontrolled hypertension, diabetes mellitus (DM), peripheral neuropathy, and infectious diseases (including viral, bacterial and parasitic infections), etc.
8. Pregnancy or lactation, or a fertility plan during the participation in this study.
9. No more than 4 weeks or no more than 5 times of t1/2 since prior investigational agents.
10. Other situations that impede the patient's participation in the study at the discretion of the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-10-30 (Estimated); Study Completion 2018-11-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Plasma Concentration [Cmax] | Day 0 - Day 21 for single dose and Day 28 - Day 63 for multiple doses
  part 1 for single dose and part 2 for multiple doses
Half life of CPGJ602 in blood [t1/2] | Day 0 - Day 21 for single dose and Day 28 - Day 63 for multiple doses
  part 1 for single dose and part 2 for multiple doses
Area Under the Curve [AUC] | Day 0 - Day 21 for single dose and Day 28 - Day 63 for multiple doses
  part 1 for single dose and part 2 for multiple doses
Incidence of Adverse Events [AEs] | Day -28 to 1 month following the last administration
  to evaluate the safety and tolerability

SECONDARY OUTCOMES:
Anti-Drug Antibody [ADA] | Day 0 to Day 63, and in the follow-up period.
  to evaluate the Immunogenicity; if the result is positive, Neutralizing Antibody [NAB] will also be assessed.
Objective Response Rate [ORR] | Day -28 - Day 63
  the rate of completely response [CR] and partial response [PR] patients
Carcinoembryonic antigen [CEA] | Day -28 - Day 63
  Tumor Marker
Cancer antigen [CA19-9] | Day -28 - Day 63
  Tumor Marker

CONTACTS AND LOCATIONS:
Overall Officials: Jianming Xu, Doctor, Principal Investigator — the Afflicated Hospital of Academy of Military Medical Sciences
Locations (1):
- Sir Run Run Shaw Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided